CLINICAL TRIAL: NCT06829849
Title: Validity of the SHD-LESS Scale in Detecting Landing Asymmetry and Its Association With Functional Status After ACL Reconstruction.
Brief Title: Validity of the SHD-LESS Scale After ACL Reconstruction
Acronym: ACL-LESS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: ACL-LESS
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: ACL Reconstruction; ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL reconstruction group: All sports patients who had a muscle evaluation at 6 to 12 months after ACLR since March 2024
  Interventions: Diagnostic Test: Landing error assessment during a SHD task using the SHD-LESS scale

INTERVENTIONS:
Diagnostic Test: Landing error assessment during a SHD task using the SHD-LESS scale — Participants will perform a 2D-camera-recorded SHD task, with the SHD-LESS scored by two sports medicine physicians. Additional tests include isokinetic muscle testing, as well as functional and psychological status assessments, following standard clinical practice.

SUMMARY:
After anterior cruciate ligament reconstruction (ACL-R), Single Hop for Distance (SHD) performance aids in decision-making, particularly for return-to-sport assessments. However, asymmetrical landing kinematics are common after ACL-R, even with symmetrical performances, and increase the risk of re-injury. To support clinical practice, several qualitative scales have been developed as valid and reliable tools for assessing landing quality. In 2022, Measson et al. adapted the Landing Error Scoring System for use during an SHD task (SHD-LESS scale) and demonstrated its reliability among healthy individuals.

The aim of this study is to test the validity of this scale after ACL-R by evaluating its ability to identify asymmetrical landing and characterize differences between the operated and uninjured limb. The second objective is to assess its association with knee muscle strength, functional status and psychological readiness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40, who have undergone a first ACL reconstruction more than 6 months ago and are being followed in a sports medicine care pathway
* Affiliated with a health insurance plan
* Information form: Non-objection to the use of data for research purposes

Exclusion Criteria:

* Previous ligament surgery of the lower limbs prior to ACL reconstruction
* Complex ligament injury (lateral ligaments, posterior cruciate ligament)
* Recent muscle injuries
* History of injury to the uninjured knee
* Pregnant woman
* Inability to perform a muscular assessment
* Postoperative complications (deep vein thrombosis, sepsis, stiffness/arthrofibrosis)
* Neurological history with residual effects or taking medication that affects balance/coordination

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All sports patients included in the sport medicine follow-up protocole with isokinetic muscular assessment at 6-12 months after ACL reconstruction surgery since March 2024 in the sports medicine department (Return To Sport Process)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Single Hop for Distance, Landing Error Scoring System (SHD-LESS) scale | One measurement during the visit at 6 to 12 months after surgery
  The LESS (Landing Error Scoring System) scale is a 13-item tool used to assess landing technique during a hop task.

SECONDARY OUTCOMES:
Strength | One measurement during the visit at 6 to 12 months after surgery
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer
ACL-RSI questionnaire (Anterior Cruciate Ligament-Return to Sport after Injury) | One measurement during the visit at 6 to 12 months after surgery
  The ACL-RSI measures the patient's understanding of his knee. It comprises 12 questions with a score of 1 to 10 for each
International Knee Documentation Committee (IKDC) score | One measurement during the visit at 6 to 12 months after surgery
  Knee level of function based on patient-reported measures from symptoms to daily activities. The IKDC score includes sections on knee symptoms (7 items), function (2 items), and sports activities (2 items), with scores ranging from 0 (lowest function, highest symptoms) to 100 (highest function, lowest symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine du sport, CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Measson MV, Ithurburn MP, Rambaud AJ. Intra-rater Reliability of a Qualitative Landing Scale for the Single-Hop Test: A Pilot Study. Int J Sports Phys Ther. 2022 Apr 1;17(3):493-500. doi: 10.26603/001c.33066. eCollection 2022. PMID 35391866
- [Background] Welling W, Benjaminse A, Seil R, Lemmink K, Gokeler A. Altered movement during single leg hop test after ACL reconstruction: implications to incorporate 2-D video movement analysis for hop tests. Knee Surg Sports Traumatol Arthrosc. 2018 Oct;26(10):3012-3019. doi: 10.1007/s00167-018-4893-7. Epub 2018 Mar 16. PMID 29549389